CLINICAL TRIAL: NCT06091501
Title: LIVING - Physical Activity in a Self-management Program Among Persons With Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other); Region Zealand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LIVING
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 2; Randomized Controlled Trial
Keywords: Diabetes self-management program; High intensity interval training
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study is designed as a parallel-group, 2-arm pragmatic RCT. The primary outcome is diabetes competences measured by The Perceived Competence in Diabetes scale (PCD) before and after 8 weeks of interventions. The trial sites are to deliver either (1) Lev Livet or (2) Lev Livet + HiiT. Within each trial site the participants will be randomly allocated (2:1) to intervention or a control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lev Livet (Experimental): The participants will receive the 9 weeks of Lev Livet intervention
  Interventions: Behavioral: Lev Livet
- Lev Livet control (No Intervention): The participants will attend 5 months of waiting list
- Lev Livet + HiiT (Experimental): The participants will receive the 9 weeks of Lev Livet intervention AND 9 weeks of HiiT training
  Interventions: Behavioral: Lev Livet
- Lev Livet + HiiT control (No Intervention): The participants will attend 5 months of waiting list

INTERVENTIONS:
Behavioral: Lev Livet — The program consists of a total of 9 sessions with a duration of two and a half to three hours for each session. In the first four sessions coping skills are taught across different chronic diseases. In this part of the program citizens suffering from different chronic diseases can participate. Citizens living with T2D then move on to four diabetes-specific sessions, followed by a ninth follow up session. The sessions are held consecutively over eight weeks. The ninth session is held three weeks after the eighth session.
  The 8 weeks supervised HIIT-protocol will be comprised of blocks of 5 x 1 min high-intensity intervals interrupted by 1 min active recovery. The HIIT intervention will progress continuously, from two weekly training sessions with two training blocks (22 minutes of training) in the first two weeks, to two weekly training sessions with four training blocks in the last four weeks of the intervention.
  Arms: Lev Livet; Lev Livet + HiiT

SUMMARY:
The goal of this pragmatic clinical trial is to evaluate two municipality-based interventions, Lev Livet (one without physical activity and one with) against no intervention in people with type 2 diabetes. The main questions it aims to answer are: • What is the additive effect of HiiT on accelerometer-measured physical activity? • Which factors that facilitate or limit the implementation of Lev Livet? • What are the health-economic implications of the intervention? Participants will participate in a disease management program with and without physical activity added. Researchers will compare with no intervention to see if Lev Livet improves diabetes self-management.

DETAILED DESCRIPTION:
Trial design The LIVING project is designed as a parallel-group, 2-arm pragmatic RCT. The trial sites are to deliver either sub study 1: Lev Livet versus a five month waiting list or sub study 2: Lev Livet + HIIT versus a five month waiting list. At the clarifying interview with a health professional in the municipality, the participants will be randomly allocated to either Lev Livet (+HIIT) or a waiting list (control group). Within each sub study, the participants will be randomly allocated (2:1) to intervention or a control group.

Participants All people living with T2D being referred from their general practitioner or a hospital to the municipality can be included in the project.

Intervention Lev Livet is a group-based program where the aim for the participant is to acquire skills to master their daily life with T2D. The program consists of 9 sessions with a duration of two and a half to three hours for each session. In the first four sessions coping skills are taught across different chronic diseases. In this part of the program citizens suffering from different chronic diseases can participate. Participants living with T2D then move on to four diabetes-specific sessions, followed by a ninth follow up session. The eight first sessions are held consecutively over eight weeks. The ninth session is held three weeks after the eighth session.

During the 8 weeks, a supervised HIIT-protocol comprising blocks of 5 x 1 min high-intensity intervals interrupted by 1 min active recovery will be added. Between each blocks, a 4 min brake will be planned where the participant can shift from an upper body exercise to a lower body exercise or vice versa. The HIIT intervention will progress continuously, from two weekly exercise sessions with two exercise blocks (22 minutes of exercise) in the first two weeks, to two weekly exercise sessions with four exercise blocks in the last four weeks of the intervention. The exercise intensity will be monitored using the Borg 15 scale. The intensity of exercise will be set to Borg 14-16 corresponding to 77-93% of maximal heart rate. In addition to the two exercise therapy sessions, the participants will be instructed to independently complete an exercise session equivalent to the exercise therapy session for that week.

Statistical analyses The primary analyses of both the primary and secondary outcomes will be based on the mean difference between individual changes from baseline to 3 months when comparing the Lev Livet intervention and control group.

Analysis will be done according to the intention-to-treat principle, meaning that all participants allocated to an active treatment group will be analysed as a member of that group regardless of their compliance with the intervention. Missing data will be imputed in the primary analysis using a multiple imputation procedure29.

The analysis will be performed using a mixed model with repeated measures. Specifically, time as a categorical covariate, randomisation status, and their interaction will be included. This will allow assessment of difference at each time point of follow-up between groups, as well as of the overall difference. Dependence of repeated observations for participants will be handled with a random effect for participant. In addition, random effects for group and municipality will be included, assuming independence between random effects at different levels (participant, group, municipality). To explore the effect of adding HIIT to the intervention, the investigators will use a mixed model as described above, but with an added interaction term between sub study 2, sub study 1 and follow-up status. Further, the effect of adding HIIT to the intervention will be explored on other outcomes conducting analysis of mediation.

Analyses of baseline equivalence between groups of intervention and control group will be performed. In order to increase precision of the outcome estimate, covariates can be included in the analyses if relevant.

Power calculation and sample size In a realistic real-world set-up, each municipality will be able to run two rounds of intervention, e.g. randomize participants into two intervention groups and two control groups. The intervention to control group ratio is estimated to be 2:1. Number of participants in each intervention group is expected to be 12 and 6 in each control group, meaning that each municipality has to randomise 36 participants. A simulation procedure was applied to estimate the power assuming a difference in change between groups of 5 and that individual changes had an SD (standard deviation) of 4. Including four municipalities in each sub study, 8 in total (288 participants in total) would yield a power of 80%.

Qualitative study on the health care professionals' perspective To gain knowledge on the implementation process of the intervention Lev Livet, and Lev Livet + HIIT, the perspectives of the providing health care professionals will be investigated13.

During the delivery of the intervention, the experiences of twenty to thirty healthcare professionals from various sites will be examined. Data collection will include participant observations30 and focus group interviews31. The following research questions will guide data collection:

* What is at stake in clinical practice when delivering the intervention?
* How do healthcare professionals perceive their relation to the patients during the intervention?
* What characterizes the health care support given to patients during the intervention? Thematic analysis32 will lead to new insight into the healthcare professional perspective during the intervention, relevant for further refinements and implementation.

Qualitative approach to explore participants' experiences Inspired by realistic evaluation33, the aim is to explore what parts of the disease management program work for whom and why. This includes an exploration of the barriers of implementing new knowledge and habits from Lev Livet into the participants' daily lives as well as the elements they have successfully implemented.

After completing Lev Livet, participants from sub study 2 in two different municipalities (n=24), will be invited for an interview. Using a semi-structured, open-ended interview methodology34, the interviews will touch upon topics such as; their daily life with diabetes, expectations before participating in Lev Livet, their experienced outcomes, motivation to participate and carry on with new habits, and being part of a group with a disease in common.

Participants in the first round of interviews will be invited for follow-up interviews four to six months later. These will focus on how the participants have managed their diabetes since Lev Livet, which habits they have or have not implemented into their daily lives and which factors play into what works in their daily setting.

Health economic evaluation As there are expectedly multiple effects of varying character, a cost consequence analysis will be performed to analyse the health economic consequences of the intervention. The costs of the Lev Livet intervention as well as the HIIT component is estimated and these costs are related to the primary and secondary outcomes collectively. When estimating the costs, a rigorous approach will be applied. This includes identifying all relevant cost components in collaboration with project participants, measuring the resources consumed using the most appropriate method for each cost component, and finally calculating the monetary value by using individual unit prices35.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T2D
* Age >=18 years
* able to speak and understand Danish
* individuals assessed fit by a health care professional to attend a diabetes self-management program

Exclusion Criteria:

* Contraindication to increasing level of physical activity assessed by the participant' general practitioner (e.g. unstable angina, uncontrolled arrhythmias or severe aortic stenosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The between group differences for change in Perceived competence in Diabetes (PCS-5) | From baseline to endpoint (month 3) and follow-up (month 5, 8 and 12)
  PCS-5 is a five 5-item scale with seven response categories from not at all true to very, true, assessing the degree to which the individual feel they can manage their diabetes. Range 7-35 with higher scores indicating higher competences in managing own diabetes.

SECONDARY OUTCOMES:
The between group differences for change in physical activity | From baseline to endpoint (month 3) and follow-up month 5
  The accelerometer-measured outcome is defined as purposeful moderate-to-vigorous physical activity in people living with T2D

CONTACTS AND LOCATIONS:
Overall Officials: Anette Andersen, Principal Investigator — Aarhus University Hospital, Denmark
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jensen JM, Sorensen KV, Stovring H, Andersen A. LIVING - protocol for a pragmatic randomized controlled trial investigating the effect of three different levels of diabetes self-management programs. Contemp Clin Trials. 2025 Jun;153:107891. doi: 10.1016/j.cct.2025.107891. Epub 2025 Mar 29. PMID 40164303